CLINICAL TRIAL: NCT04021550
Title: Combined Treatment of Angiotensin Receptor Blocker and Antioxidant Supplementation as a Novel Adjunctive Therapy for 24-hour Blood Pressure Improvement in Obstructive Sleep Apnea
Brief Title: Improving 24-hour Blood Pressure in Obstructive Sleep Apnea
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Covid-19 Pandemic prevented this study from beginning
Sponsor: University of British Columbia (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Glen Foster, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H18-03130
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Telmisartan; Alpha-Lipoic Acid; Continuous Positive Airway Pressure; 24-hour blood pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Telmisartan; Thioctic Acid; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Treatment (Experimental): Subjects will be given 80 mg/day Telmisartan + 600 mg/day Alpha-Lipoic Acid. Subjects will also be prescribed CPAP therapy by their physician. Subjects will be instructed to use their CPAP device according to their physician's guidelines.
  Interventions: Device: Continuous Positive Airway Pressure CPAP; Drug: Telmisartan 80mg; Dietary Supplement: Alpha-Lipoic Acid 600mg
- Placebo Control (Placebo Comparator): Subjects will be given placebo capsules. Subjects will also be prescribed CPAP therapy by their physician. Subjects will be instructed to use their CPAP device according to their physician's guidelines.
  Interventions: Device: Continuous Positive Airway Pressure CPAP; Other: Microcrystalline Cellulose

INTERVENTIONS:
Device: Continuous Positive Airway Pressure CPAP — All subjects will be advised to use their continuous positive airway pressure (CPAP) in accordance to their physician's guidelines.
Drug: Telmisartan 80mg — Subjects in this group will receive 80mg/day of Telmisartan (an angiotensin receptor blocker). Treatments will be administered in pre-packaged blister packages. Subjects will take Telmisartan once per day for 6 weeks.
  Arms: Combined Treatment
Dietary Supplement: Alpha-Lipoic Acid 600mg — Subjects in this group will receive 600mg/day of Alpha-Lipoic Acid (an antioxidant). Treatments will be administered in pre-packaged blister packages. Subjects will take Alpha-Lipoic Acid once per day for 6 weeks.
  Arms: Combined Treatment
Other: Microcrystalline Cellulose — Subjects in this group will receive two capsules of Microcrystalline Cellulose (placebo). Treatments will be administered in pre-packaged blister packages. Subjects will take placebo pills once per day for 6 weeks.
  Arms: Placebo Control

SUMMARY:
This study examines the combined effects of an angiotensin receptor blocker (ARB), antioxidant supplementation, and continuous positive airway pressure (CPAP) therapy on the lowering of 24-hour blood pressure in persons with moderate to severe Obstructive Sleep Apnea (OSA). All participants will undergo CPAP therapy as prescribed by their doctor; however, half of the participants will receive the combined ARB and antioxidant treatment while the other half of the participants will receive a placebo.

DETAILED DESCRIPTION:
OSA is a sleep disorder characterized by repetitive collapses (apneas) or partial collapses (hypopneas) of the upper airway. These airway obstructions result in intermittent reductions in arterial oxygen saturation (hypoxia), which causes a reflexive increase in sympathetic activation and systemic vasoconstriction. Resumption of breathing results in transient surges in blood pressure (BP) that can reach as high as 240/130 mm/Hg.

OSA effects up to 24% of the adult population and evidence suggests a causal relationship between OSA and cardiovascular disease (CVD) development. While the exact mechanisms are unknown, data from animal and human models suggest that exposure to chronic intermittent hypoxia (IH) plays a significant role in the pathogenesis of cardiovascular comorbidity. Persons with OSA exhibit increased daytime sympathetic activity, markers of oxidative stress, and vasoactive hormones, particularly angiotensin II, that contribute to systemic vasoconstriction. These factors contribute to early endothelial dysfunction and contribute to sustained elevations in BP.

While CPAP is the gold standard OSA treatment, adherence rates are low and evidence suggests that treatment does not reduce the rates of CVD in large population-based studies.

Telmisartan is a receptor blocker for angiotensin II and not only has BP lowering effects, but also has unique anti-inflammatory properties and beneficial influences on endothelial function. The addition of an antioxidant supplement may increase the reactive oxygen species scavenging capacity and, in combination with ARB treatment, may provide more robust effects on BP in persons with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Apnea/Hypopnea Index (AHI) greater than/equal to 15 events per hour of sleep
* No prior use of CPAP
* Body mass index less than 30kg/m2
* Does not take ARBs or angiotensin converting enzyme inhibitors for blood pressure control
* Females of childbearing potential on an effective or highly effective means of contraception

Exclusion Criteria:

* Prescribed and/or taking the following medications: diuretics (including potassium-sparing diuretics), Digoxin, lithium salts, and/or nonsteroidal anti-inflammatory drugs
* Over the counter supplements that affect the cardiovascular system, such as fish oils, vitamins, or other antioxidants
* History of heart failure
* History of myocardial infarction
* History of coronary artery disease
* History of stroke
* History of diabetes mellitus
* History of impaired renal function
* History of chronic obstructive pulmonary disease
* History of asthma
* History of central sleep apnea
* Smoked within the past year
* Hypotensive (Systolic blood pressure (SBP) <90 mmHg and diastolic blood pressure (DBP) <60 mmHg)
* Females who do not have a means of contraception, are pregnant, planning to become pregnant, and/or are breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour blood pressure | Change from baseline of 24-hour systolic, diastolic, and mean arterial blood pressure at 6 weeks
  Systolic, diastolic, and mean arterial blood pressure (mmHg)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frampton JE. Telmisartan: a review of its use in cardiovascular disease prevention. Drugs. 2011 Apr 16;71(6):651-77. doi: 10.2165/11206710-000000000-00000. PMID 21504246
- [Background] Khayat RN, Varadharaj S, Porter K, Sow A, Jarjoura D, Gavrilin MA, Zweier JL. Angiotensin Receptor Expression and Vascular Endothelial Dysfunction in Obstructive Sleep Apnea. Am J Hypertens. 2018 Feb 9;31(3):355-361. doi: 10.1093/ajh/hpx174. PMID 29036393
- [Background] Khayat R, Patt B, Hayes D Jr. Obstructive sleep apnea: the new cardiovascular disease. Part I: Obstructive sleep apnea and the pathogenesis of vascular disease. Heart Fail Rev. 2009 Sep;14(3):143-53. doi: 10.1007/s10741-008-9112-z. Epub 2008 Sep 20. PMID 18807180
- [Background] Rotenberg BW, Murariu D, Pang KP. Trends in CPAP adherence over twenty years of data collection: a flattened curve. J Otolaryngol Head Neck Surg. 2016 Aug 19;45(1):43. doi: 10.1186/s40463-016-0156-0. PMID 27542595
- [Background] Pepin JL, Tamisier R, Barone-Rochette G, Launois SH, Levy P, Baguet JP. Comparison of continuous positive airway pressure and valsartan in hypertensive patients with sleep apnea. Am J Respir Crit Care Med. 2010 Oct 1;182(7):954-60. doi: 10.1164/rccm.200912-1803OC. Epub 2010 Jun 3. PMID 20522795